CLINICAL TRIAL: NCT03822000
Title: Risk Factors and Complications Contributing to Mortality in Elderly Patients With Fall-Induced Femoral Fracture: A Cross-sectional Analysis Based on Trauma Registered Data
Brief Title: Risk Factors and Complications Contributing to Mortality in Elderly Patients With Fall-Induced Femoral Fracture
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CDRPG8H0011-2
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Femoral Fractures
Keywords: femur fracture; trauma; fall; elderly; mortality; respiratory complication
MeSH Terms: conditions — Femoral Fractures; Wounds and Injuries | interventions — Death Domain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Patients with Femoral Fracture: Elderly patients with fall-induced femoral fracture. Patients were categorized into two groups: death (n = 42) and survival (n = 2,365).
  Interventions: Other: Survival; Other: Death

INTERVENTIONS:
Other: Survival — Elderly patients with fall-induced femoral fracture who were survived.
Other: Death — Elderly patients with fall-induced femoral fracture who were dead.

SUMMARY:
This study aimed to identify the risk factors and complications associated with mortality in elderly patients with femoral fracture after a fall from the ground level.

DETAILED DESCRIPTION:
This retrospective study reviewed data pertaining to elderly patients aged ≥ 65 years who were admitted into a Level I trauma center, between January 1, 2009 and December 31, 2017. Multivariate logistic regression analysis was performed to identify independent effects of univariate predictive variables on the occurrence of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a fall from ≥1 m as well as those for whom incomplete data were available.

Exclusion Criteria:

* those patients with a fall from ≥1 m
* patients with incompleted data

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This retrospective study reviewed data from 27,462 trauma patients registered between January 1, 2009 and December 31, 2016. The inclusion criteria were age ≥65 years and hospitalization for the treatment of femoral fracture following a fall from standing height level (<1 m). This study excluded those patients with a fall from ≥1 m as well as those for whom incomplete data were available.
Sampling Method: Probability Sample
Enrollment: 2407 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Mortality | up tp 2 months
  Mortality was used as the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan